CLINICAL TRIAL: NCT00266825
Title: Kansas University DHA Outcome Study (KUDOS)
Brief Title: DHA Supplementation and Pregnancy Outcome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Susan Carlson, PhD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Susan Carlson, PhD, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10186; R01HD047315 (NIH)
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Pregnancy
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA capsules (Experimental): DHA capsules
  Interventions: Drug: DHA
- Placebo capsules (Placebo Comparator): Placebo capsule
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Drug: DHA — 600 mg DHA
  Other Names: docosahexaenoic acid
  Arms: DHA capsules
Other: Placebo capsule — Placebo capsule
  Arms: Placebo capsules

SUMMARY:
The purpose of the study is to determine if increasing DHA intake during pregnancy can increase gestation duration and enhance infant and childhood outcomes related to visual acuity, stereoacuity, attention, and distractibility.

DETAILED DESCRIPTION:
Although numerous trials show benefits of postnatal DHA supplementation for visual acuity and others show benefits for cognitive function and/or attention, studies of increased DHA exposure during fetal life are needed, especially in the US. Women in the US consume low amounts of DHA compared to other world populations, and this likely means less DHA transfer to the fetus than in many other populations. Prenatal DHA exposure may be more important than postnatal exposure, because animal studies show critical windows for brain DHA accumulation in relation to effects on neurotransmitters such as serotonin, dopamine and GABA.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant 8-20 wks at enrollment
* single fetus
* BMI <40

Exclusion Criteria:

* diabetes (Type I, ii, GDM)
* hypertension (primary, PIH, preeclampsia/eclampsia)

Ages: 16 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 350 (Actual)
Dates: Start 2006-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Carlson, PhD, Principal Investigator — University of Kansas Medical Center; John Colombo, PhD, Principal Investigator — University of Kansas
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Truman Medical Center, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Carlson SE, Colombo J, Gajewski BJ, Gustafson KM, Mundy D, Yeast J, Georgieff MK, Markley LA, Kerling EH, Shaddy DJ. DHA supplementation and pregnancy outcomes. Am J Clin Nutr. 2013 Apr;97(4):808-15. doi: 10.3945/ajcn.112.050021. Epub 2013 Feb 20. PMID 23426033
- [Result] Ozias MK, Kerling EH, Christifano DN, Scholtz SA, Colombo J, Carlson SE. Typical prenatal vitamin D supplement intake does not prevent decrease of plasma 25-hydroxyvitamin D at birth. J Am Coll Nutr. 2014;33(5):394-9. doi: 10.1080/07315724.2013.879843. Epub 2014 Oct 10. PMID 25302772
- [Result] Scholtz SA, Kerling EH, Shaddy DJ, Li S, Thodosoff JM, Colombo J, Carlson SE. Docosahexaenoic acid (DHA) supplementation in pregnancy differentially modulates arachidonic acid and DHA status across FADS genotypes in pregnancy. Prostaglandins Leukot Essent Fatty Acids. 2015 Mar;94:29-33. doi: 10.1016/j.plefa.2014.10.008. Epub 2014 Nov 7. PMID 25500337
- [Derived] Colombo J, Shaddy DJ, Gustafson K, Gajewski BJ, Thodosoff JM, Kerling E, Carlson SE. The Kansas University DHA Outcomes Study (KUDOS) clinical trial: long-term behavioral follow-up of the effects of prenatal DHA supplementation. Am J Clin Nutr. 2019 May 1;109(5):1380-1392. doi: 10.1093/ajcn/nqz018. PMID 31004139
- [Derived] Carlson SE, Gajewski BJ, Alhayek S, Colombo J, Kerling EH, Gustafson KM. Dose-response relationship between docosahexaenoic acid (DHA) intake and lower rates of early preterm birth, low birth weight and very low birth weight. Prostaglandins Leukot Essent Fatty Acids. 2018 Nov;138:1-5. doi: 10.1016/j.plefa.2018.09.002. Epub 2018 Sep 20. PMID 30392575
- [Derived] Lepping RJ, Honea RA, Martin LE, Liao K, Choi IY, Lee P, Papa VB, Brooks WM, Shaddy DJ, Carlson SE, Colombo J, Gustafson KM. Long-chain polyunsaturated fatty acid supplementation in the first year of life affects brain function, structure, and metabolism at age nine years. Dev Psychobiol. 2019 Jan;61(1):5-16. doi: 10.1002/dev.21780. Epub 2018 Oct 11. PMID 30311214
- [Derived] Hidaka BH, Thodosoff JM, Kerling EH, Hull HR, Colombo J, Carlson SE. Intrauterine DHA exposure and child body composition at 5 y: exploratory analysis of a randomized controlled trial of prenatal DHA supplementation. Am J Clin Nutr. 2018 Jan 1;107(1):35-42. doi: 10.1093/ajcn/nqx007. PMID 29381793
- [Derived] Hidaka BH, Kerling EH, Thodosoff JM, Sullivan DK, Colombo J, Carlson SE. Dietary patterns of early childhood and maternal socioeconomic status in a unique prospective sample from a randomized controlled trial of Prenatal DHA Supplementation. BMC Pediatr. 2016 Nov 25;16(1):191. doi: 10.1186/s12887-016-0729-0. PMID 27884184
- [Derived] Yelland LN, Gajewski BJ, Colombo J, Gibson RA, Makrides M, Carlson SE. Predicting the effect of maternal docosahexaenoic acid (DHA) supplementation to reduce early preterm birth in Australia and the United States using results of within country randomized controlled trials. Prostaglandins Leukot Essent Fatty Acids. 2016 Sep;112:44-9. doi: 10.1016/j.plefa.2016.08.007. Epub 2016 Aug 17. PMID 27637340
- [Derived] Shireman TI, Kerling EH, Gajewski BJ, Colombo J, Carlson SE. Docosahexaenoic acid supplementation (DHA) and the return on investment for pregnancy outcomes. Prostaglandins Leukot Essent Fatty Acids. 2016 Aug;111:8-10. doi: 10.1016/j.plefa.2016.05.008. Epub 2016 May 13. PMID 27499448
- [Derived] Colombo J, Gustafson KM, Gajewski BJ, Shaddy DJ, Kerling EH, Thodosoff JM, Doty T, Brez CC, Carlson SE. Prenatal DHA supplementation and infant attention. Pediatr Res. 2016 Nov;80(5):656-662. doi: 10.1038/pr.2016.134. Epub 2016 Jun 30. PMID 27362506
- [Derived] Colombo J, Carlson SE, Cheatham CL, Shaddy DJ, Kerling EH, Thodosoff JM, Gustafson KM, Brez C. Long-term effects of LCPUFA supplementation on childhood cognitive outcomes. Am J Clin Nutr. 2013 Aug;98(2):403-12. doi: 10.3945/ajcn.112.040766. Epub 2013 Jun 26. PMID 23803884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from the Kansas City metro area. Enrollment occurred between January 2006 and November 2009.
Groups:
- DHA Supplement: DHA capsule
  DHA: 600 mg DHA
Period: Enrolled and Allocated Intervention
Arm/Group | Placebo Capsule | DHA Supplement
Started | 172 | 178
Completed | 172 | 178
Not Completed | 0 | 0
Period: Completed Follow-Up
Arm/Group | Placebo Capsule | DHA Supplement
Started | 172 | 178
Completed | 147 | 154
Not Completed | 25 | 24
Not completed — Lost to Follow-up | 14 | 19
Not completed — Withdrawal by Subject | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Capsule | DHA Supplement | Total
Number analyzed (Participants) | 172 | 178 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (4.7) | 25.3 (4.9) | 25.0 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 178 | 350
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Race of mother
  participants
    Black | 79 | 66 | 145
    Not Black | 93 | 112 | 205
Race/Ethnicity, Customized [Number; unit: participants] — Ethnicity of mother
  participants
    Hispanic | 14 | 14 | 28
    Not Hispanic | 158 | 164 | 322
Region of Enrollment [Number; unit: participants]
  United States | 172 | 178 | 350
Gestation at Enrollment [Mean (Standard Deviation); unit: days] | 99.6 (26.1) | 102.9 (25.3) | 101.3 (25.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Total Fatty Acids by Weight
Description: Measure of RBC-phospholipid-DHA at Birth
Time Frame: at time of birth
Population: The effect of DHA supplementation on study primary outcomes was determined for black and non-black subjects separately. Researchers did not compare outcomes between black and non-black subjects to determine whether they were statistically different. For measures reporting black and non-black results, there were 184 non-black and 117 black subjects.
Measure: Mean (Standard Deviation); unit: percentage of fatty acid
Arm/Group | Placebo Capsule | DHA Supplement
Number analyzed (Participants) | 147 | 154
percentage of fatty acid
  All Subjects | 4.7 (1.3) | 7.3 (2.2)
  Not Black Subjects (n=93, 112)) | 4.8 (1.3) | 7.8 (2.1)
  Black Subjects (n=79, 66) | 4.7 (1.3) | 6.2 (2.0)

2. Secondary Outcome: Ponderal Index
Description: Ponderal index calculated with formula Weight (g)/length (cm)^3 * 100. It a measure of leanness of a person and is calculated as a relationship between mass and height. Commonly used in pediatrics.
Time Frame: at time of birth
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Capsule | DHA Supplement
Number analyzed (Participants) | 147 | 154
units on a scale | 2.7 (0.4) | 2.7 (0.3)

3. Primary Outcome: Gestational Age
Description: Gestational age of babies at time of birth in days
Time Frame: at time of birth
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Capsule | DHA Supplement
Number analyzed (Participants) | 147 | 154
days
  All Subjects | 272.8 (17.0) | 275.7 (11.2)
  Not Black Subjects (n=93,112) | 273.8 (14.0) | 275.9 (9.9)
  Black Subjects (n=79,66) | 271.4 (20.3) | 275.2 (13.3)

4. Primary Outcome: Birth Weight
Description: Weight of baby at birth
Time Frame: at time of birth
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Placebo Capsule | DHA Supplement
Number analyzed (Participants) | 147 | 154
grams
  All Subjects | 3187 (602) | 3359 (524)
  Not Black Subjects (n=93,112) | 3282 (529) | 3489 (456)
  Black Subjects (n=79,66) | 3060 (671) | 3110 (559)

5. Primary Outcome: Birth Length
Description: Length of baby at birth
Time Frame: at time of birth
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Placebo Capsule | DHA Supplement
Number analyzed (Participants) | 147 | 154
centimeters
  All Subjects | 49.0 (3.4) | 49.7 (2.7)
  Not Black Subjects (n=93,112) | 49.2 (2.9) | 50.0 (2.6)
  Black Subjects (n=79,66) | 48.6 (4.0) | 49.0 (2.7)

6. Secondary Outcome: Gender of Babies
Time Frame: at time of birth
Measure: Number; unit: percentage of babies
Arm/Group | Placebo Capsule | DHA Supplement
Number analyzed (Participants) | 147 | 154
percentage of babies
  Male | 54 | 49
  Female | 46 | 51

7. Secondary Outcome: Cord RBC-phospholipid-DHA
Description: Percentage of total fatty acids by weight in cord RBC
Time Frame: at time of birth
Measure: Mean (Standard Deviation); unit: percentage of cord RBC
Arm/Group | Placebo Capsule | DHA Supplement
Number analyzed (Participants) | 147 | 154
percentage of cord RBC | 5.9 (1.4) | 7.3 (1.8)

8. Secondary Outcome: Head Circumference
Description: Measure of circumference of baby's head in centimeters at time of birth.
Time Frame: at time of birth
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Placebo Capsule | DHA Supplement
Number analyzed (Participants) | 147 | 154
centimeters | 33.7 (2.0) | 34.2 (1.7)

9. Secondary Outcome: Preterm Births
Description: Percentage of births occurring at less than 37 weeks of gestation.
Time Frame: births before week 37 of gestation
Measure: Number; unit: percentage of births
Arm/Group | Placebo Capsule | DHA Supplement
Number analyzed (Participants) | 147 | 154
percentage of births | 8.8 | 7.8

ADVERSE EVENTS:
Time Frame: Researchers followed the mother for 30 days post-partum and the infant from birth to 18 months. Typical follow-up stops 30 days after the end of the intervention. Researchers collected information on each from their medical records.
Groups:
- Placebo Capsule - Mother: Placebo capsule
  Placebo capsule: Placebo capsule
- Placebo Capsule - Infant: Infants born from Mothers in the Placebo capsule group
- DHA Capsule - Mother: DHA capsule
  DHA: 600 mg DHA
- DHA Capsule - Infant: Infants born from Mothers in the DHA capsule group
Arm/Group | Placebo Capsule - Mother | Placebo Capsule - Infant | DHA Capsule - Mother | DHA Capsule - Infant
Serious Adverse Events (participants affected / at risk) | 18/147 | 31/147 | 18/154 | 26/154
Other Adverse Events (participants affected / at risk) | 0/147 | 0/147 | 0/154 | 0/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Capsule - Mother (N=147) | Placebo Capsule - Infant (N=147) | DHA Capsule - Mother (N=154) | DHA Capsule - Infant (N=154)
Hospitalization or miscarriage (Pregnancy, puerperium and perinatal conditions) | 18 (18) | 0/0 (0) | 18 (18) | 0/0 (0)
Hospitalization and death (Pregnancy, puerperium and perinatal conditions) | 0/0 (0) | 31 (31) | 0/0 (0) | 26 (26)
Congenital anomalies (Congenital, familial and genetic disorders) | 0/0 (0) | 2 (2) | 0/0 (0) | 5 (5)
Postpartum hospitalization (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0/0 (0) | 1 (1) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes